CLINICAL TRIAL: NCT02091466
Title: Pre-warming With Thermal Gown Prevents Maternal Hypothermia in Elective Cesarean Section
Brief Title: Pre-warming Prevents Hypothermia in Elective Cesarean Section
Acronym: hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Caio Gracco De Bernardis, PhD, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 388/08 - FCMSCSP
Record Dates: First submitted 2014-03-13; First posted 2014-03-19 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2014-09

CONDITIONS: Hypothermia
Keywords: Hypothermia; Perioperative Care; Anesthesia; Spinal; Rewarming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-warming (Active Comparator): The intervention is to warm patients before the anesthesia procedure in experimental groups
  Interventions: Device: pre-warming
- Control (No Intervention): Patients received no active warming before the anesthesia procedure in control groups

INTERVENTIONS:
Device: pre-warming — warming patients 30 minutes prior to anesthesia
  Arms: Pre-warming

SUMMARY:
Background: Hypothermia is common during general and regional anesthesia even when active warming measures are taken. The existing literature shows that, in pregnant patients, the use of forced air-warming during cesarean section under spinal anesthesia does not prevent maternal hypothermia. Therefore, this study aimed to establish the efficacy of a pre-warming system, initiated 30 minutes before the onset of spinal anesthesia and during surgery, in pregnant women subjected to elective cesarean delivery.

Methods: Forty healthy pregnant patients undergoing elective cesarean section with spinal anesthesia were allocated to the control group (Gcont, n = 20), without the use of a thermal gown, and to the gown group (Ggown, n = 20), with the use of a thermal gown in the preoperative care unit, 30 minutes before spinal anesthesia installation and during surgery. After the anesthesia, the thermal gown was moved from the regular position and placed over the chest and upper limbs, as an upper body blanket, and maintained throughout the study. The following variables were observed: preoperative and operative room temperature, hemoglobin saturation, heart rate, arterial pressure, tympanic temperature in the preoperative care unit room (baseline) and at 0, 15, 30, 45 and 60 minutes after spinal anesthesia. Repeated Measure ANCOVA compared temperatures of each group, adjusted for baseline values.

DETAILED DESCRIPTION:
Introduction Body temperature decreasing following the onset of general or regional anesthesia is caused by a core-to-peripheral redistribution of heat, as demonstrated by several previous studies. Perioperative hypothermia and its complications have been widely studied in patients subjected to non-obstetric surgery; however, literature on the obstetric population is rare, although the incidence of intraoperative shivering can be as high as 60% in these patients. A previous study based on the use of forced air-warming unit during the preoperative and intraoperative periods in patients subjected to cesarean delivery observed a lower incidence of hypothermia and shivering in patients given epidural anesthesia when compared to those given spinal anesthesia.

The forced air system is by far the most commonly used intraoperative warming approach and has an admirable safety record. However, the problem with blanket-forced air warming, circulating-water garments, or water mattresses is that it is impossible to change their position on the bed, which can be uncomfortable, especially if the patient is waiting in a sitting position.

The Bair Paws Gown® presents an air warming system that provides patient-controlled comfort warming in the pre and postoperative setting. The same gown offers effective clinical warming during surgery involving the head, neck, knees or extremities. The air-warming flows through the gown, from knees to head or from head to knees, and allows the patient to be seated with gown covering the area between knees and neck.

Therefore, we designed a study to establish the efficacy of a pre-warming system that keeps the garment throughout the perioperative period, without interruption, initiated 30 minutes before the induction of spinal anesthesia for elective cesarean delivery. The aim of this study was to test the hypothesis that active warming 30 minutes before spinal anesthesia should better prevent a fall in pregnant body temperature. A secondary goal evaluated the incidence of shivering, as well as thermal comfort during the procedure.

Methods After obtaining Institutional Review Board approval (record 388/08) and written informed consent from patients, 40 healthy ASA physical status I or II pregnant women presenting for scheduled cesarean delivery under spinal anesthesia were enrolled in this prospective, randomized study.

Randomization (1:1) was based on a random computer generated code that was maintained in sequentially numbered opaque envelopes.

Eligible participants were pregnant women between 18 and 40 years of age, with singleton pregnancy and gestation longer than 37 weeks, scheduled for elective cesarean section. Patients with fever and/or infectious conditions, a familial history of potential malignant hyperthermia, body mass index (BMI) values below 18.5 kg.cm-2 or above 36 kg.cm-2, thyroid disorders, dysautonomia, Raynaud's syndrome, and those in labor were excluded.

Participants remained seated in the preoperative care unit until they were allocated to one of the following groups: control group (Gcont n = 20), in which surgery was performed without the use of a thermal gown, or gown group (Ggown n = 20), in which surgery was performed while the patients were covered with a thermal gown (Bair Paws Standard Warming Gown 810 model with a Bair Hugger, model 850 warming unit) with forced-air flow at 40ºC in the preoperative care unit 30 minutes before the spinal anesthesia. When the patients were transferred to the operative room, the warming gown was switched off for the gown group; however, the gown was maintained in place and, when the pregnant women arrived in operative room, the system was switched back on and the gown was moved to the anterior part of the body, covering chest and upper limbs as an upper body blanket, which was maintained until the end of surgery.

In the operative room, a venous cannula was inserted into the forearm, and an infusion of Ringer's lactate solution fluids at 37ºC was initiated. Spinal anesthesia was administered using 10 mg of hyperbaric bupivacaine, combined with 10 µg of fentanyl and 80 µg of morphine. Puncture was performed at level L1-L2 or L2-L3 of the lumbar vertebra, and surgery began when the sensory blockage reached a level between the T4 and T6 thoracic vertebra, as established by the loss of sensitivity to needle pricks. Intraoperative hydration used 500 ml of 40ºC Ringer's lactate solution before fetal extraction and 800 µg metaraminol was provided via slow infusion or 400 µg was delivered as an IV bolus whenever the arterial pressure decreased by more than 25% of the baseline value. Following fetal extraction but before the end of surgery, 1,000 ml of Ringer's lactate solution with 20 IU of oxytocin was infused.

Demographic variables included age, weight, height and BMI. Patients were monitored with hemoglobin peripheral saturation (SpO2), heart rate (HR), noninvasive systolic arterial pressure (SAP) and diastolic arterial pressure (DAP). The tympanic temperature was measured by means of a digital thermometer (Techline Model TS 201, Sao Paulo, SP, Brazil) Ambient temperature was maintained approximately at 22ºC according to wall thermostat (ABNT NBR 7256 - Brazilian regulatory and normalization Agency).

All data were assessed at baseline, 30 minutes before induction of spinal anesthesia; T0 (immediately after the spinal anesthesia); and T15, T30, T45, and T60 (15, 30, 45, and 60 minutes following the onset of spinal anesthesia, respectively).

In addition, postoperative data were assessed during the admission to the post-anesthesia care unit (PACU). Shivering was evaluated according to Wrench's scale that uses: 0 - no shivering; 1 - one or more symptoms of piloerection, peripheral vasoconstriction, and peripheral cyanosis without any other cause and without visible muscular activity; 2 - visible muscular activity confined to one muscle group; 3 - visible muscular activity in more than one muscle group; and 4 - gross muscular activity involving the entire body. Thermal discomfort according to Horn's verbal numerical scale: 0 - worst imaginable cold, 100 - insufferably hot and adverse effects during the immediate postoperative period were also registered. Moreover, patients received 12.5-25 mg meperidine whenever their shivering scores were equal to or greater than three.

Sample size was calculated to be 20 participants to ensure that a difference of 0.5ºC could be detected at significance level of 5%, with a statistical power of 80%, assuming the standard deviation of differences to be 0.5ºC.

Data are presented as mean and standard deviation or median and interquartile interval (25-75) according to tested distribution (Shapiro-Wilk test). Analysis of covariance for repeated measures (ANCOVA), adjusted for baseline values, compared tympanic temperatures between the groups. Statistical significance was established at p < 0.05, and the statistical analysis was performed using SPSS (Statistical Package for the Social Sciences) software version 20.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* between 18 and 40 years of age
* singleton pregnancy
* gestation longer than 37 weeks
* elective cesarean section

Exclusion Criteria:

* fever and/or infectious conditions
* familial history of potential malignant hyperthermia
* body mass index (BMI) values below 18.5 kg.cm-2 or above 36 kg.cm-2
* thyroid disorders, dysautonomia, Raynaud's syndrome
* patient in labor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Caio G De Bernardis, M.D. Ph.D, Principal Investigator — Irmandade Santa Casa deMisericórdia de São Paulo
Locations (1):
- Irmandade Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were pregnant women between 18 and 40 years of age, with singleton pregnancy and gestation longer than 37 weeks, scheduled for elective cesarean section, between March 18, 2010 and July 17, 2010 - assisted at the Obstetric Clinic of Santa Casa de Misericórdia de São Paulo.
Pre-assignment Details: Patients with fever (peripheral temperature > 37.8 Celsius) and/or infectious conditions, familial history of potential malignant hyperthermia, body mass index (BMI) values below 18.5 Kg.m-2 or above 36 Kg.m-2, thyroid disorders, dysautonomia, Raynaud's syndrome, and those in labor were excluded.
Groups:
- Pre-warming: patients were under heating system in experimental groups
  heating system pre-warming: warming 30 minutes prior to anesthesia
- Control: patients were under passive heating in control groups before anesthesia
Period: Overall Study
Arm/Group | Pre-warming | Control
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-warming; Control: Eligible participants were pregnant women between 18 and 40 years of age, with singleton pregnancy and gestation longer than 37 weeks, scheduled for elective cesarean section
- Total: Total of all reporting groups
Arm/Group | Pre-warming | Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (5.9) | 28.4 (6.0) | 28.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Maternal Hypothermia
Description: Hypothermia was measured by means of tympanic temperatures.
Time Frame: 60 minutes
Population: Sample size was calculated to be 20 subjects in each group to ensure that a difference of 0.5ºC at 60 minutes could be detected at significance level of 5% with a statistical power of 90%, assuming the standard deviation of differences to be 0.5ºC, considering a temperature below 36.0ºC could be considered hypothermia
Measure: Mean (Standard Deviation); unit: Centigrades
Groups:
- Pre-warming: Patients were covered with a thermal gown (Bair Paws Standard Warming Gown 810 model with a Bair Hugger, model 850 warming unit) with forced-air flow at 40ºC in the preoperative care unit 30 minutes before the spinal anesthesia.
- Control: Patients remained without the use of a thermal gown,
Arm/Group | Pre-warming | Control
Number analyzed (Participants) | 20 | 20
Centigrades
  baseline | 36.6 (0.3) | 36.4 (0.4)
  time zero | 36.5 (0.3) | 36.3 (0.3)
  15 minutes | 36.4 (0.3) | 35.9 (0.4)
  30 minutes | 36.2 (0.3) | 35.7 (0.4)
  45 minutes | 36.2 (0.3) | 35.6 (0.3)
  60 minutes | 36.1 (0.2) | 35.4 (0.4)
Statistical Analysis 1: Comparison: Pre-warming vs Control; Analysis of covariance for repeated measures (ANCOVA), adjusted for baseline values, compared tympanic temperatures between the groups. Statistical significance was established at p < 0.05, and the statistical analysis was performed using SPSS (Statistical Package for the Social Sciences) software version 20; Test type: Superiority or Other; p < 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: Up to 6 hours
Description: shivering during Post-Anesthesia Care Unit
Arm/Group | Pre-warming | Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No